CLINICAL TRIAL: NCT04930367
Title: CombinADO: a Cluster-randomized Controlled Trial to Compare the Efficacy, Uptake, Feasibility and Acceptability of the CombinADO Strategy Versus Optimized Standard of Care on Viral Suppression, ART Adherence and Retention in HIV Care Among Adolescents and Young Adults Living with HIV Ages 10-24yrs in Nampula Province, Mozambique
Brief Title: CombinADO: Evaluation of an Intervention Aimed At Improving HIV Outcomes Among Adolescents and Young Adults Living with HIV in Mozambique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Cape Town (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Senior Research Director, ICAP, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAT5971; 4UH3HD096926-03 (NIH)
Record Dates: First submitted 2021-06-05; First posted 2021-06-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV
Keywords: HIV; Adolescents; Mozambique; ART adherence; Viral suppression
MeSH Terms: interventions — Health Personnel; Seroconversion

STUDY DESIGN:
Intervention Model Description: A cluster-randomized trial to compare the effectiveness of the CombinADO strategy versus optimized standard of care (SOC) on viral suppression, ART adherence and retention in HIV care among AYAHIV ages 10-24yrs attending participating health facilities. Clinics are the units of intervention allocation and randomization. The control condition will be implemented at all facilities (n=12) participating in the trial. The enhanced intervention condition will be superadded to this at a randomly selected half (n=6) of facilities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Standard of Care (Active Comparator): To be implemented at all 12 clinic sites, includes a set of interventions aimed at optimizing the national standard of care (billboards/posters and radio shows, healthcare worker training, one-stop adolescent and youth friendly services, information/motivation walls, pill containers and tools to be used by clinic staff during clinical visits)
  Interventions: Behavioral: Radio Ads; Behavioral: Community Sensitization Campaign; Behavioral: Informational Posters; Behavioral: Motivation Walls; Other: Pill Container; Other: CombinADO-specific training for healthcare workers; Other: One Stop Shop Model of Care; Other: Treatment Toolkit; Other: Self-reflection Kit
- CombinADO Strategy (Experimental): To be implemented at 6 randomly selected clinic sites, includes all interventions in the "Enhanced Standard of Care" arm plus five additional intervention components, including 1) Mental health screening and linkage to adolescent-focused mental health support, 2) peer navigation support, 3) an informational video, 4) peer support groups for AYAHIV and 5) support groups for caregivers of AYAHIV
  Interventions: Behavioral: Radio Ads; Behavioral: Community Sensitization Campaign; Behavioral: Informational Posters; Behavioral: Motivation Walls; Other: Pill Container; Other: CombinADO-specific training for healthcare workers; Other: One Stop Shop Model of Care; Other: Treatment Toolkit; Other: Self-reflection Kit; Behavioral: Peer Support; Behavioral: Informational and motivational Video; Behavioral: Support groups- caregivers of adolescents and young adults living with HIV; Behavioral: Support groups- adolescents and young adults living with HIV; Behavioral: Mental health screening and linkage to adolescent-focused mental health support

INTERVENTIONS:
Behavioral: Radio Ads — Engaging radio mini shows that address community stigma and medical literacy through busting common myths with humor and building empathy with heartfelt storytelling.
Behavioral: Community Sensitization Campaign — Large-scale, infographic billboards and posters located in public areas and secondary schools to address stigma, medical literacy and promote community support for AYAHIV.
Behavioral: Informational Posters — Large-scale, infographic posters located in clinic waiting areas to normalize HIV and build confidence in treatment.
Behavioral: Motivation Walls — Interactive, patient-generated posters located in the consultation room where patients can post words and phrases about themselves and their futures.
Other: Pill Container — A discreet pill container to support ART adherence.
Other: CombinADO-specific training for healthcare workers — Comprehensive in-service training for healthcare workers focused on the needs of adolescents and young adults living with HIV
Other: One Stop Shop Model of Care — Model of care that allows adolescents and young adults living with HIV to access a complete set of services, including HIV care, in one central location.
Other: Treatment Toolkit — A guide to clinic visits and discussions on ART and viral load monitoring to help healthcare workers better communicate with patients.
Other: Self-reflection Kit — A simple handout for healthcare workers to help patients reflect on their ART progress and understand the concept of viral load as a measure of ART success.
Behavioral: Peer Support — Peer exposure to examples of adolescents and young adults openly living with HIV (AYAHIV) and; opportunities to share their experiences with HIV in one-on-one interactions with other AYAHIV during clinic visits.
  Arms: CombinADO Strategy
Behavioral: Informational and motivational Video — An informational and motivational video that in simple language with engaging graphics that a) demystifies and simplifies HIV, ART, and viral load and; b) emphasizes that people can live long, healthy lives.
  Arms: CombinADO Strategy
Behavioral: Support groups- caregivers of adolescents and young adults living with HIV — A learning, support, and empowerment group for caregivers of adolescents and young adults living with HIV (AYAHIV). Through monthly gatherings, the program aims to foster confidence, and equip caregivers with strategies to support AYAHIV adherence journey.
  Arms: CombinADO Strategy
Behavioral: Support groups- adolescents and young adults living with HIV — A peer-to-peer learning, support, and empowerment group to address loss of hope and improve medical literacy. Through biweekly gatherings, the program aims to foster belonging and confidence, equipping young people and caregivers with strategies to navigate the adherence journey.
  Arms: CombinADO Strategy
Behavioral: Mental health screening and linkage to adolescent-focused mental health support — HCWs will be trained in the use of a brief mental health screening tool focusing on depression, anxiety, and post-traumatic stress disorder. Mental health service providers at each facility will be trained and supported to provide diagnostic and mental health support to youth with positive screens who agree to further evaluation.
  Arms: CombinADO Strategy

SUMMARY:
This is a cluster-randomized trial designed to compare the effectiveness of the CombinADO strategy versus optimized standard of care (SOC) on viral suppression, antiretroviral therapy (ART) adherence and retention in HIV care among adolescents living with HIV (ALHIV) ages 10 to 24 years attending participating health facilities. Clinics are the units of intervention allocation and randomization. The control condition will be implemented at all facilities (n=12) participating in the trial. The enhanced intervention condition will be superadded to this at a randomly selected half (n=6) of facilities. The goal of this study is to learn whether an enhanced, tailored intervention helps AYAHIV do better with their HIV care (take their medications, stay in care) than the usual care that they receive.

DETAILED DESCRIPTION:
HIV burden among adolescents and young people worldwide is substantial, with an estimated 1.7 million adolescents aged 10-19 years living with HIV in 2019, and 460,000 adolescents aged 15-24 newly infected reported in the same year. Adolescent girls continue to be disproportionately affected, accounting for 56% of new infections worldwide. With increased availability of antiretroviral therapy (ART), pediatric mortality has decreased and healthcare workers (HCW) are now challenged to meet the complex needs of the large number of surviving youth who must cope with HIV as a chronic, highly stigmatized, and transmittable illness. There are 1.8 billion people between ages 10 and 24 and it is projected that the number of people <20 years will double by 2030. In sub-Saharan Africa (SSA), youth aged 10-24 years comprise 30-35% of the countries' population. Failure to prevent new HIV infections among adolescents will result in increased numbers of adolescents and young adults living with HIV (AYAHIV) who will strain health and social service systems as they transition to adulthood.

ELIGIBILITY:
Adolescents and young adults living with HIV (AYAHIV):

Inclusion Criteria:

1. HIV-positive, per medical records and confirmed by health facility staff
2. Age 10 to 24 years
3. Registered as a patient at study site
4. Aware of HIV+ status
5. Provision of signed and dated informed consent form
6. For adolescents under 18 years of age, informed assent and parental informed consent to participate in the study
7. Stated willingness to comply with all study procedures

Exclusion Criteria:

1. Has an acute medical condition requiring immediate medical care

Caregivers of AYAHIV:

Inclusion Criteria:

1. Age 18 years and older
2. Attending a caregiver-specific support group
3. Willingness to be audio-recorded

Healthcare Workers (HCW) and Key Informants (KI):

Inclusion Criteria:

1. Age 18 years and older
2. Involved in the provision, management, or oversight of adolescent-focused HIV services at the 12 specified study sites
3. Willingness to be audio-recorded

For all study participants (AYAHIV, caregivers, HCW and KI):

Exclusion Criteria:

Any other condition, including but not limited to alcohol or substance abuse and uncontrolled medical condition and/or allergies, that, in the opinion of the study team, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives would make the patient unsuitable for the study or unable/unwilling to comply with the study requirements.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1715 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Proportion of adolescents and young people living with HIV (AYAHIV) with viral suppression (Viral load <50 copies/ml) | 12 months post intervention implementation
  Viral suppression among AYAHIV at intervention versus control sites

SECONDARY OUTCOMES:
Proportion of eligible adolescents and young people living with HIV (AYAHIV) attending clinic in a 90 day window from end of intervention implementation, as assessed at 12 months post intervention. | 12 months post intervention implementation
  Retention in HIV care & treatment among AYAHIV at intervention versus control sites
Self-reported adherence measured using 3-item adherence scale (mean score) | 12 months post intervention implementation
  Self-reported ART adherence among adolescents and young people living with HIV at intervention versus control sites will be measured using a three-item adherence scale. The three items include (1) an assessment of the number of days with missed ART doses in the preceding 30 days [0-30 days]; (2) a scale rating of how good a job you did taking your medicines in the preceding 30 days (never/rarely/sometimes/usually/almost always/always) and (3) a scale rating of how often you took your medicines the way you were supposed to in the preceding 30 days (very poor/poor/fair/good/very good/ excellent).
  For analyses using raw scores, item responses for the three adherence items will be linearly transformed to a 0-100 scale with zero being the worst adherence, and 100 representing perfect adherence. The mean of the three scores are then taken to get an equally weight aggregate scale score. An overall mean from the scores from all participants will be reported.
Proportion of participants with detectable antiretroviral (ARV) on dried blood spot (DBS) specimen | 12 months post intervention implementation
  ART adherence among among adolescents and young people living with HIV (AYAHIV) at intervention versus control sites, ARV levels

CONTACTS AND LOCATIONS:
Overall Officials: Elaine J Abrams, MD, Principal Investigator — ICAP at Columbia University
Locations (12):
- Mozambique (12):
  - Cs 1 de Maio, Nampula
  - Cs 25 Setembro, Nampula
  - Cs Alua, Nampula
  - Cs Anexo Psi, Nampula
  - Cs Malema, Nampula
  - Cs Muhala Expansao, Nampula
  - Cs n1 Nacala Porto, Nampula
  - Cs Nametil, Nampula
  - Cs Namialo, Nampula
  - Cs Namicopo, Nampula
  - HG Marere, Nampula
  - HR Angoche, Nampula

IPD SHARING:
Plan to Share IPD: Yes
As required by study funder, de-identified, archived data will be transmitted to and stored at NICHD's Data and Specimen Hub (DASH) for use by other researchers including those outside of the study. Permission to transmit data to DASH will be included in the informed consent signed by all study participants. This data will only be shared after the end of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within one year after end of the study
Access Criteria: When the study is completed, access to study data will be provided through NICHD's DASH repository. Researchers seeking to access data stored in DASH will need to follow pre-specified requirements around data access requests.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Derived] Mogoba P, Falcao J, Tolla T, Zerbe A, De Gusmao EP, Myer L, Abrams EJ. A qualitative evaluation of stakeholder perspectives on the implementation of HIV services within adolescent and youth-friendly services for the youth in Nampula, Mozambique. BMC Health Serv Res. 2025 Sep 30;25(1):1229. doi: 10.1186/s12913-025-13414-0. PMID 41029606
- [Derived] Mogoba P, Lesosky M, Mukonda EE, Zerbe A, Falcao J, Zandamela R, Myer L, Abrams EJ. Positive attitudes toward adoption of a multi-component intervention strategy aimed at improving HIV outcomes among adolescents and young people in Nampula, Mozambique: perspectives of HIV care providers. BMC Health Serv Res. 2023 Jun 6;23(1):582. doi: 10.1186/s12913-023-09630-1. PMID 37280638
- [Derived] Mogoba P, Lesosky M, Zerbe A, Falcao J, Mellins CA, Desmond C, Arnaldo C, Kapogiannis B, Myer L, Abrams EJ. The CombinADO study to assess the impact of a combination intervention strategy on viral suppression, antiretroviral therapy adherence, and retention in HIV care among adolescents and young people living with HIV: protocol for a cluster-randomized controlled trial. Trials. 2021 Dec 27;22(1):956. doi: 10.1186/s13063-021-05943-w. PMID 34961567